CLINICAL TRIAL: NCT06272019
Title: Alternative Application Methods of Pre-procedural Povidone Iodine Mouthrinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannakorn Sriarj, Assistant professor, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HREC-DCU 2023-074
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: The Retention of Iodine in Saliva Over the Time; The Comparison of Iodine in Saliva Between Gargle and Swab

STUDY DESIGN:
Intervention Model Description: the participant will use iodine gargle in 2 method
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gargle method (Experimental): the participant will use 0.2% iodine gargle with gargle method by hold in mouth 30 second and gargle 30 seconds after that spit out
  Interventions: Other: Iodine gargle
- Swab method (Experimental): the participant will use 0.2 iodine gargle with swab method by the researcher apply on mouth 1 minute without spit out
  Interventions: Other: Iodine gargle

INTERVENTIONS:
Other: Iodine gargle — Iodine gargle 0.2 %

SUMMARY:
To compare the iodine remaining in saliva between gargle method and swab method

DETAILED DESCRIPTION:
separate the participant in 2 groups group 1 use iodine gargle with gargle method, after 48 hours use iodine gargle with swab method group 2 use iodine gargle with swab method, after 48 hours use iodine gargle with gargle method The researcher will collect saliva before use iodine gargle and after use at time 0, 5, 10, 20, 30, 60, 120 minutes

ELIGIBILITY:
Inclusion Criteria:

* Thai people
* no underlying disease, no pregnant
* at least 24 teeth
* No use iodine gargle
* No allergy to iodine and seafood
* No orthodontic and prosthetic treatment
* No ulcer and edentulous area
* Saliva flow rate in male (0.57+-0.3 ml/minute), in woman (0.41+-0.27 ml/minute)
* PI score lower than 0.6 (Green and vermillion index)

Exclusion Criteria:

* treatment orthodontic or prosthetic treatment currently
* Allergy to iodine between reach
* Can not participate

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
The rate of retention of iodine in saliva | 0, 5, 10, 20, 30, 60 and 120 minutes
  The retention of iodine in saliva after get the gargle (show in percentage)
The comparison of the retention of iodine between gargle and swab | 0, 5, 10, 20, 30, 60 and 120 minutes
  The comparison of rate of retention of iodine in saliva between gargle and swab (show in percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Wannakorn Sriar, Principal Investigator — Faculty of Dentistry, Chulalongkorn University
Locations (1):
- Faculty of Dentistry, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tabatabaeizadeh SA. Airborne transmission of COVID-19 and the role of face mask to prevent it: a systematic review and meta-analysis. Eur J Med Res. 2021 Jan 2;26(1):1. doi: 10.1186/s40001-020-00475-6. PMID 33388089
- [Background] Hu B, Guo H, Zhou P, Shi ZL. Characteristics of SARS-CoV-2 and COVID-19. Nat Rev Microbiol. 2021 Mar;19(3):141-154. doi: 10.1038/s41579-020-00459-7. Epub 2020 Oct 6. PMID 33024307
- [Background] Zou X, Chen K, Zou J, Han P, Hao J, Han Z. Single-cell RNA-seq data analysis on the receptor ACE2 expression reveals the potential risk of different human organs vulnerable to 2019-nCoV infection. Front Med. 2020 Apr;14(2):185-192. doi: 10.1007/s11684-020-0754-0. Epub 2020 Mar 12. PMID 32170560
- [Background] Chen L, Zhao J, Peng J, Li X, Deng X, Geng Z, Shen Z, Guo F, Zhang Q, Jin Y, Wang L, Wang S. Detection of SARS-CoV-2 in saliva and characterization of oral symptoms in COVID-19 patients. Cell Prolif. 2020 Dec;53(12):e12923. doi: 10.1111/cpr.12923. Epub 2020 Oct 19. PMID 33073910
- [Background] Xu H, Zhong L, Deng J, Peng J, Dan H, Zeng X, Li T, Chen Q. High expression of ACE2 receptor of 2019-nCoV on the epithelial cells of oral mucosa. Int J Oral Sci. 2020 Feb 24;12(1):8. doi: 10.1038/s41368-020-0074-x. PMID 32094336
- [Background] Okui T, Matsuda Y, Karino M, Hideshima K, Kanno T. Oral Mucosa Could Be an Infectious Target of SARS-CoV-2. Healthcare (Basel). 2021 Aug 19;9(8):1068. doi: 10.3390/healthcare9081068. PMID 34442205
- [Background] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Background] Lippi G, Mattiuzzi C, Bovo C, Plebani M. Current laboratory diagnostics of coronavirus disease 2019 (COVID-19). Acta Biomed. 2020 May 11;91(2):137-145. doi: 10.23750/abm.v91i2.9548. PMID 32420937
- [Background] Ge ZY, Yang LM, Xia JJ, Fu XH, Zhang YZ. Possible aerosol transmission of COVID-19 and special precautions in dentistry. J Zhejiang Univ Sci B. 2020 May;21(5):361-368. doi: 10.1631/jzus.B2010010. Epub 2020 Mar 16. PMID 32425001
- [Background] Jamal M, Shah M, Almarzooqi SH, Aber H, Khawaja S, El Abed R, Alkhatib Z, Samaranayake LP. Overview of transnational recommendations for COVID-19 transmission control in dental care settings. Oral Dis. 2021 Apr;27 Suppl 3(Suppl 3):655-664. doi: 10.1111/odi.13431. Epub 2020 Jun 3. PMID 32428372
- [Background] Peng X, Xu X, Li Y, Cheng L, Zhou X, Ren B. Transmission routes of 2019-nCoV and controls in dental practice. Int J Oral Sci. 2020 Mar 3;12(1):9. doi: 10.1038/s41368-020-0075-9. PMID 32127517
- [Background] Cochran MA, Miller CH, Sheldrake MA. The efficacy of the rubber dam as a barrier to the spread of microorganisms during dental treatment. J Am Dent Assoc. 1989 Jul;119(1):141-4. doi: 10.14219/jada.archive.1989.0131. PMID 2760346
- [Background] Samaranayake LP, Reid J, Evans D. The efficacy of rubber dam isolation in reducing atmospheric bacterial contamination. ASDC J Dent Child. 1989 Nov-Dec;56(6):442-4. PMID 2681303
- [Background] Samaranayake LP, Peiris M. Severe acute respiratory syndrome and dentistry: a retrospective view. J Am Dent Assoc. 2004 Sep;135(9):1292-302. doi: 10.14219/jada.archive.2004.0405. PMID 15493394
- [Background] Kariwa H, Fujii N, Takashima I. Inactivation of SARS coronavirus by means of povidone-iodine, physical conditions and chemical reagents. Dermatology. 2006;212 Suppl 1(Suppl 1):119-23. doi: 10.1159/000089211. PMID 16490989
- [Background] Eggers M, Koburger-Janssen T, Eickmann M, Zorn J. In Vitro Bactericidal and Virucidal Efficacy of Povidone-Iodine Gargle/Mouthwash Against Respiratory and Oral Tract Pathogens. Infect Dis Ther. 2018 Jun;7(2):249-259. doi: 10.1007/s40121-018-0200-7. Epub 2018 Apr 9. PMID 29633177
- [Background] Ather A, Patel B, Ruparel NB, Diogenes A, Hargreaves KM. Coronavirus Disease 19 (COVID-19): Implications for Clinical Dental Care. J Endod. 2020 May;46(5):584-595. doi: 10.1016/j.joen.2020.03.008. Epub 2020 Apr 6. PMID 32273156
- [Background] Bidra AS, Pelletier JS, Westover JB, Frank S, Brown SM, Tessema B. Comparison of In Vitro Inactivation of SARS CoV-2 with Hydrogen Peroxide and Povidone-Iodine Oral Antiseptic Rinses. J Prosthodont. 2020 Aug;29(7):599-603. doi: 10.1111/jopr.13220. Epub 2020 Jul 24. PMID 32608097
- [Background] Martinez Lamas L, Diz Dios P, Perez Rodriguez MT, Del Campo Perez V, Cabrera Alvargonzalez JJ, Lopez Dominguez AM, Fernandez Feijoo J, Diniz Freitas M, Limeres Posse J. Is povidone iodine mouthwash effective against SARS-CoV-2? First in vivo tests. Oral Dis. 2022 Apr;28 Suppl 1(Suppl 1):908-911. doi: 10.1111/odi.13526. Epub 2020 Jul 29. No abstract available. PMID 32615642
- [Background] Reis INR, do Amaral GCLS, Mendoza AAH, das Gracas YT, Mendes-Correa MC, Romito GA, Pannuti CM. Can preprocedural mouthrinses reduce SARS-CoV-2 load in dental aerosols? Med Hypotheses. 2021 Jan;146:110436. doi: 10.1016/j.mehy.2020.110436. Epub 2020 Nov 27. PMID 33288313
- [Background] Rattanawiboon C, Chaweewannakorn C, Saisakphong T, Kasevayuth K, Trairatvorakul C. Effective Fluoride Mouthwash Delivery Methods as an Alternative to Rinsing. Nurs Res. 2016 Jan-Feb;65(1):68-75. doi: 10.1097/NNR.0000000000000131. PMID 26657482
- See also: interim guidance for minimizing risk of COVID-19transmission — https://snlg.iss.it/wp-content/uploads/2020/04/ADA_COVID_Int_Guidance_Treat_Pts.pdf
- See also: Thai dental guideline — https://www.royalthaident.org/content/13